CLINICAL TRIAL: NCT00739388
Title: 5-Azacytidine to Treat Acute Myeloid Leukemia in Elderly or Frail Patients Not Suitable for Intensive Chemotherapy. A Multicenter Phase II Trial.
Brief Title: Azacitidine in Treating Patients With Newly Diagnosed Previously Untreated or Secondary Acute Myeloid Leukemia Who Are Unsuitable For Intensive Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 30/07; SWS-SAKK-30/07; CDR0000612029
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm: 5-azacytidine (Experimental): 5-azacytidine 100 mg/m2/day s.c. on days 1-5 of a 28-day cycle.
  Interventions: Drug: azacytidine

INTERVENTIONS:
Drug: azacytidine — 100 mg/m2/day s.c. on days 1-5 of a 28-day cycle
  Other Names: Azacitidine; 5-azacytidine; Vidaza

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well azacitidine works in treating patients with acute myeloid leukemia who are unsuitable for treatment with intensive chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of azacitidine in patients with newly diagnosed or untreated acute myeloid leukemia who are unsuitable for induction type chemotherapy because of age or relevant comorbidities.

Secondary

* To evaluate survival and adverse events.

OUTLINE: This is a multicenter study.

Patients receive azacitidine subcutaneously on days 1-5. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * De novo acute myeloid leukemia (AML)
  * AML secondary to prior hematological disease or cytotoxic treatment
* Newly diagnosed or untreated disease
* At least 20% blasts in the blood or bone marrow or extramedullary disease
* Must be considered unsuitable for intensive chemotherapy due to ≥ 1 of the following:

  * High age or frail for the biologic age
  * Relevant comorbidities
  * Unwilling to undergo intensive chemotherapy
* No chronic myelogenous leukemia or acute promyelocytic leukemia

PATIENT CHARACTERISTICS:

* WHO performance status 0-3
* Bilirubin ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* AST ≤ 2.5 times ULN
* Serum creatinine ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* Patient compliance and geographic proximity allow proper staging and follow-up
* No NYHA class III-IV heart failure or relevant cardiac arrhythmia
* No active hematological/oncological disease other than AML
* No psychiatric disorder precluding understanding of information on trial related topics or giving informed consent
* No serious underlying medical condition in the judgment of the investigator, which could impair the ability of the patient to participate in the trial, including but not limited to, any of the following:

  * Active autoimmune disease
  * Uncontrolled diabetes
  * Active uncontrolled infection
  * HIV infection
  * Active chronic hepatitis B or C infection
* No known allergy or hypersensitivity to azacitidine or mannitol

PRIOR CONCURRENT THERAPY:

* No prior treatment for AML
* No prior azacitidine or decitabine
* No other concurrent experimental or investigational drugs or anticancer therapy
* More than 30 days since participation in another clinical trial
* No concurrent growth factors for use in afebrile and asymptomatic patients except to treat neutropenic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Best response (complete or partial response) | within 6 months

SECONDARY OUTCOMES:
Time to response | is defined as the time from trial registration until the date the criteria for either CR or PR are first met
Response duration | is defined as the time from the date when the criteria for either CR or PR were first met until the date of relapse or death from any cause.
Best response status | within 6 months
Time to hematological improvement (HI) | is calculated for patients with HI and is defined as the time from trial registration until the date the criteria for HI are first met.
Duration of HI | is defined as the time from the date when the criteria for HI were first met until the date of relapse or death from any cause.
Event-free survival | is defined as the time from trial registration until progression, relapse or death from any cause, whichever occurs first.
Overall survival | is defined as the time from trial registration until death from any cause.
Adverse events according to NCI CTCAE v3.0 | according to NCI CTCAE v3.0
Adjusted hospitalization time | is defined as the time (nights) spent in hospital as a proportion of treatment duration (days).

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Passweg, Prof, Study Chair — Hopitaux Universitaires de Geneve; Sabine Blum, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (11):
- Switzerland (11):
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital, Luzerne, Luzerne
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hopitaux Universitaires de Geneve, Thonex-Geneve
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Passweg JR, Pabst T, Blum S, Bargetzi M, Li Q, Heim D, Stussi G, Gregor M, Leoncini L, Meyer-Monard S, Brauchli P, Chalandon Y; Swiss Group for Clinical Cancer Research (SAKK). Azacytidine for acute myeloid leukemia in elderly or frail patients: a phase II trial (SAKK 30/07). Leuk Lymphoma. 2014 Jan;55(1):87-91. doi: 10.3109/10428194.2013.790540. Epub 2013 May 2. PMID 23547838